CLINICAL TRIAL: NCT05194228
Title: Exemplar: Determining the Best Practices for EMA Studies
Acronym: Exemplar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 13684
Record Dates: First submitted 2021-11-10; First posted 2022-01-18 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Ecological Momentary Assessment Best Practices
Keywords: Ecological Momentary Assessment; Health Behavior; Smartphone Application
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into 1 of 32 conditions in a 2x2x2x2x2 design (i.e., number of questions per EMA survey [15 vs. 25] x number of EMAs per day [2 vs. 4] x EMA prompting schedule [random vs. fixed times]) x payment type [per EMA vs. based on percentage of EMAs completed] x order of EMA item question types [i.e., slider type first 2 weeks vs. Likert-type questions first 2 weeks]).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (32):
- Group 1 (Experimental): $1 Payment per EMA 2 EMAs per day 15 questions per EMA Fixed schedule Slider first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 2 (Experimental): $1 Payment per EMA 2 EMAs per day 15 questions per EMA Fixed schedule Likert first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 3 (Experimental): $1 Payment per EMA 2 EMAs per day 15 questions per EMA Random schedule Slider first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 4 (Experimental): $1 Payment per EMA 2 EMAs per day 15 questions per EMA Random schedule Likert first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 5 (Experimental): $1 Payment per EMA 2 EMAs per day 25 questions per EMA Fixed schedule Slider first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 6 (Experimental): $1 Payment per EMA 2 EMAs per day 25 questions per EMA Fixed schedule Likert first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 7 (Experimental): $1 Payment per EMA 2 EMAs per day 25 questions per EMA Random schedule Slider first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 8 (Experimental): $1 Payment per EMA 2 EMAs per day 25 questions per EMA Random schedule Likert first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 9 (Experimental): $1 Payment per EMA 4 EMAs per day 15 questions per EMA Fixed schedule Slider first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 10 (Experimental): $1 Payment per EMA 4 EMAs per day 15 questions per EMA Fixed schedule Likert first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 11 (Experimental): $1 Payment per EMA 4 EMAs per day 15 questions per EMA Random schedule Slider first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 12 (Experimental): $1 Payment per EMA 4 EMAs per day 15 questions per EMA Random schedule Likert first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 13 (Experimental): $1 Payment per EMA 4 EMAs per day 25 questions per EMA Fixed schedule Slider first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 14 (Experimental): $1 Payment per EMA 4 EMAs per day 25 questions per EMA Fixed schedule Likert first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 15 (Experimental): $1 Payment per EMA 4 EMAs per day 25 questions per EMA Random schedule Slider first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 16 (Experimental): $1 Payment per EMA 4 EMAs per day 25 questions per EMA Random schedule Likert first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 17 (Experimental): Payment by % EMAs 2 EMAs per day 15 questions per EMA Fixed schedule Slider first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 18 (Experimental): Payment by % EMAs 2 EMAs per day 15 questions per EMA Fixed schedule Likert first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 19 (Experimental): Payment by % EMAs 2 EMAs per day 15 questions per EMA Random schedule Slider first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 20 (Experimental): Payment by % EMAs 2 EMAs per day 15 questions per EMA Random schedule Likert first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 21 (Experimental): Payment by % EMAs 2 EMAs per day 25 questions per EMA Fixed schedule Slider first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 22 (Experimental): Payment by % EMAs 2 EMAs per day 25 questions per EMA Fixed schedule Likert first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 23 (Experimental): Payment by % EMAs 2 EMAs per day 25 questions per EMA Random schedule Slider first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 24 (Experimental): Payment by % EMAs 2 EMAs per day 25 questions per EMA Random schedule Likert first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 25 (Experimental): Payment by % EMAs 4 EMAs per day 15 questions per EMA Fixed schedule Slider first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 26 (Experimental): Payment by % EMAs 4 EMAs per day 15 questions per EMA Fixed schedule Likert first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 27 (Experimental): Payment by % EMAs 4 EMAs per day 15 questions per EMA Random schedule Slider first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 28 (Experimental): Payment by % EMAs 4 EMAs per day 15 questions per EMA Random schedule Likert first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 29 (Experimental): Payment by % EMAs 4 EMAs per day 25 questions per EMA Fixed schedule Slider first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 30 (Experimental): Payment by % EMAs 4 EMAs per day 25 questions per EMA Fixed schedule Likert first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 31 (Experimental): Payment by % EMAs 4 EMAs per day 25 questions per EMA Random schedule Slider first
  Interventions: Behavioral: Ecologial Momentary Assessment settings
- Group 32 (Experimental): Payment by % EMAs 4 EMAs per day 25 questions per EMA Random schedule Likert first
  Interventions: Behavioral: Ecologial Momentary Assessment settings

INTERVENTIONS:
Behavioral: Ecologial Momentary Assessment settings — Various settings for ecological momentary assessments

SUMMARY:
Ecological momentary assessment (EMA) is a measurement methodology that utilizes the repeated collection of real-time data on participants' behavior and experience in their natural environment. While EMA allows researchers to gain valuable insights into dynamic behavioral processes, the need for frequent self-report can be burdensome and disruptive to participants. Compliance with EMA protocols is important for accurate, unbiased sampling, yet there is no "gold standard" for EMA study design. In the present study, the investigators aim to use a factorial design to identify the optimal components, or combinations of components, for achieving the highest compliance rates for smartphone-based ecological momentary assessments (EMAs). Participants will be randomized into 1 of 32 conditions in a 2x2x2x2x2 design (i.e., number of questions per EMA survey [15 vs. 25] x number of EMAs per day [2 vs. 4] x EMA prompting schedule [random vs. fixed times]) x payment type [per EMA vs. based on percentage of EMAs completed] x order of EMA item question types [i.e., slider type first 2 weeks vs. Likert-type questions first 2 weeks]). All participants will complete EMAs for 4 weeks. The effect of each factor on EMA compliance will be examined, as well as the effects of interactions on EMA compliance. The investigators will also examine within and between-subjects factors that influence response rates, and 2) contextual features such as environment and mood that may be associated with better compliance and participant engagement. The results of this study will have broad applications for developing best practices guidelines for future studies utilizing EMA methodologies.

DETAILED DESCRIPTION:
Ecological momentary assessment (EMA) is a measurement methodology that utilizes the repeated collection of real-time data on participants' behavior and experience in their natural environment. EMA has been used in behavioral science for years, including research examining the environmental and psychological antecedents of cigarette smoking, substance use disorders, anxiety, eating, and sleep. EMA sampling strategies are typically time-based or event-based. Time-based sampling is solicited based on a schedule; for example, a daily diary prompted every day at the same time, or at random intervals (e.g., every 3-4 hours) each day. In contrast, event- based sampling is centered around a pre-defined event and is typically initiated by the participant. For example, a participant may be asked to initiate an assessment every time the participant smokes a cigarette.

Several studies have examined the impact of EMA study design features on participant compliance. In a recent meta-analysis of compliance with EMA protocols among substance users, there was no evidence that compliance rates were associated with prompt frequency, length of assessment period, or reimbursement. Another study using a pooled dataset of 10 EMA studies found that compliance declined across days, and varied significantly depending on the time of day. In a meta-analysis of EMA studies in mental health research, a higher number of EMAs per day were associated with lower compliance, however the number of days was not. While these studies provide preliminary guidance regarding EMA study design, their results are unfortunately inconsistent, and the varied reporting across studies with respect to the definition of compliance, study design elements, and study populations make it difficult to clearly derive best practice guidelines for EMA design.

In the present study, the investigators use a factorial design to identify the optimal components, or combinations of components, for achieving the highest compliance rates for smartphone-based ecological momentary assessments (EMAs). In addition, the investigators will explore the association between EMA design features and participant compliance/response rates. A factorial design is ideal for exploring these research questions because it is statistically more efficient, as this type of design needs fewer participants to answer questions about each experimental factor of interest.6 In this study, participants will be randomized into 1 of 32 conditions (i.e., number of questions per EMA survey x number of EMAs per day x EMA prompting schedule x EMA item type x payment type) to explore:

1. both within and between-subjects factors that influence response rates, and
2. contextual features such as environment and mood that may be associated with better compliance and participant engagement. The results of this study will have broad applications for developing best practice guidelines for future studies utilizing EMA methodologies.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Demonstrate > 6th grade English literacy level
* Possess an active Android smartphone that is compatible with the Insight (TM) platform with a data plan and an operating system version 6.0 or higher
* Agree to install the study smartphone application onto their personal phone
* Agree to complete EMAs prompted by and completed through the study smartphone application

Exclusion Criteria:

* Under 18 years of age
* Demonstrates < 6th grade English literacy level
* Does not possess an active Android smartphone that is compatible with the Insight (TM) platform with a data plan and an operating system version 6.0 or higher
* Does not agree to install the study smartphone application onto their personal phone
* Does not agree to complete EMAs prompted by and completed through the study smartphone application

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Proportion of assigned daily smartphone surveys that are completed. | through study completion for each participant, 28 days
  Proportion of daily smartphone surveys completed will vary based upon group assignment.

SECONDARY OUTCOMES:
Number of minutes required to complete the smartphone-based surveys. | through study completion for each participant, 28 days
  Time to complete smartphone based surveys will vary based upon group assignment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stone, A. A., & Shiffman, S. (1994). Ecological momentary assessment (EMA) in behavorial medicine. Annals of Behavioral Medicine, 16(3), 199-202. https://doi.org/10.1093/abm/16.3.199
- [Background] Shiffman S, Stone AA, Hufford MR. Ecological momentary assessment. Annu Rev Clin Psychol. 2008;4:1-32. doi: 10.1146/annurev.clinpsy.3.022806.091415. PMID 18509902
- [Background] Jones A, Remmerswaal D, Verveer I, Robinson E, Franken IHA, Wen CKF, Field M. Compliance with ecological momentary assessment protocols in substance users: a meta-analysis. Addiction. 2019 Apr;114(4):609-619. doi: 10.1111/add.14503. Epub 2018 Dec 21. PMID 30461120
- [Background] Rintala A, Wampers M, Myin-Germeys I, Viechtbauer W. Response compliance and predictors thereof in studies using the experience sampling method. Psychol Assess. 2019 Feb;31(2):226-235. doi: 10.1037/pas0000662. Epub 2018 Nov 5. PMID 30394762
- [Background] Vachon H, Viechtbauer W, Rintala A, Myin-Germeys I. Compliance and Retention With the Experience Sampling Method Over the Continuum of Severe Mental Disorders: Meta-Analysis and Recommendations. J Med Internet Res. 2019 Dec 6;21(12):e14475. doi: 10.2196/14475. PMID 31808748
- [Background] Fletcher DJ, Lewis SM, Matthews JN. Factorial designs for crossover clinical trials. Stat Med. 1990 Oct;9(10):1121-9. doi: 10.1002/sim.4780091002. PMID 2247713
- [Derived] Kezbers KM, Robertson MC, Hebert ET, Montgomery A, Businelle MS. Detecting Deception and Ensuring Data Integrity in a Nationwide mHealth Randomized Controlled Trial: Factorial Design Survey Study. J Med Internet Res. 2025 Jan 28;27:e66384. doi: 10.2196/66384. PMID 39874573
- [Derived] Businelle MS, Hebert ET, Shi D, Benson L, Kezbers KM, Tonkin S, Piper ME, Qian T. Investigating Best Practices for Ecological Momentary Assessment: Nationwide Factorial Experiment. J Med Internet Res. 2024 Aug 12;26:e50275. doi: 10.2196/50275. PMID 39133915